CLINICAL TRIAL: NCT04968301
Title: A Cross-sectional Study: the Development of the Hip Joint Was Studied by Measuring the Anatomical Circumference of the Capsular Muscle of the Iliac Joint With Ultrasound Doppler
Brief Title: Cross-sectional Study of Ultrasonic Diagnosis of Iliac Joint Capsule Muscle
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Cui Ligang, Chief Physician, Peking University Third Hospital
Other Study IDs: M2019122
Record Dates: First submitted 2021-07-02; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-06

CONDITIONS: Femoroacetabular Impingement; Hip Developmental Dysplasia
MeSH Terms: conditions — Femoracetabular Impingement; Developmental Dysplasia of the Hip | interventions — Ultrasonography, Doppler

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- hip developmental dysplasia group: patients with developmental dysplasia of hip
  Interventions: Device: ultrasound Doppler
- femoroacetabular impingement group: patients with femoroacetabular impingement
  Interventions: Device: ultrasound Doppler
- control group: healthy volunteers
  Interventions: Device: ultrasound Doppler

INTERVENTIONS:
Device: ultrasound Doppler — A cross-sectional study:the development of the hip joint was studied by measuring the anatomical circumference of the capsular muscle of the iliac joint with ultrasound Doppler

SUMMARY:
In order to investigate the relationship between the iliac joint capsular muscle and the development of the hip joint, this study used ultrasound Doppler to measure the anatomical circumference of the iliac joint capsular muscle to explore the relationship

DETAILED DESCRIPTION:
In order to investigate the relationship between the iliac joint capsular muscle and the development of the hip joint, this study used ultrasound Doppler to measure the anatomical circumference of the iliac joint capsular muscle to explore the relationship.Ultrasound was used to compare the size of the iliac joint cystic muscle in the three groups: patients with developmental dysplasia of the hip (DDH), patients with Pincer type femoral hip impingement, and normal control group. The shear wave velocity and shear modulus of the iliac joint capsular muscle of three groups were compared to compare the degree of fat infiltration in muscle.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 20 years;
* Clinically suspected of DDH or Pincer and underwent surgery
* Understand and sign the informed consent

Exclusion Criteria:

* Leggcalve´-Perthes disease
* Muscle diseases
* Hip development disorder
* History of progressive osteoarthritis
* History of hip surgery
* History of arthritis of the hip joint
* With pacemaker or metal in the body

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who were admitted to the sports medicine outpatient department of Peking University Third Hospital for hip surgery and volunteers recruited as control group，including 40 patients with developmental dysplasia of the hip 40 femoroacetabular impingement patients and 40 healthy volunteers as the control group.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Parameter of ultraphonic results | Ultraphonic was conducted when patients were included in the study from March to October, 2019
  The anatomical circumference of the capsular muscle of the iliac joint was measured by ultrasound Doppler，including the dimensional ultrasonic gram and shear wave elasticity diagram

CONTACTS AND LOCATIONS:
Overall Officials: Ligang Cui, Principal Investigator — Peking University Third Hospital
Locations (1):
- Department of Ultrasound Diagnosis, Peking University Third Hospital, Beijing, Beijing Municipality, China